CLINICAL TRIAL: NCT05069428
Title: Delirium Reduction With Ramelteon
Acronym: DREAM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centennial Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Johnson MD, MD, Centennial Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-438
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — ramelteon

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ramelteon (Experimental): ramelteon 8 mg crushed tablet daily at 20:30
  Interventions: Drug: Ramelteon 8mg
- placebo (Placebo Comparator): placebo powder equivalent grams at 20:30
  Interventions: Drug: Ramelteon 8mg

INTERVENTIONS:
Drug: Ramelteon 8mg — administered crushed, orally at 20:30

SUMMARY:
The overall purpose of this study is to identify a medication that might treat and/or prevent delirium in intensive care unit (ICU). Currently, there is no proven medical therapy for prevention or treatment of delirium. Ramelteon is a medication approved for insomnia. We hypothesize that ramelteon may help regulate the day/night cycle and decrease ICU delirium.

DETAILED DESCRIPTION:
Melatonin is an endogenous hormone that regulates the sleep-wake cycle along with several other physiological functions. It is reported that melatonin secretion may be impaired in ICU patients, and there is some question whether this may be a contributing factor to delirium occurrence. Ramelteon is a melatonin agonist with three to six times increased affinity for MT1 and MT2 receptors versus melatonin. It is FDA approved for the treatment of insomnia, and some studies suggested some benefit with ramelteon for delirium prevention. There is limited prospective research data assessing the efficacy of ramelteon for delirium treatment. The goal of this study therefore is to assess the efficacy of ramelteon versus placebo on the prevention and treatment of delirium in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Medical or surgical ICU patient
* Ability to take oral or nasogastric tube within 48 hours of admission to ICU
* Expected ICU length of stay and life expectancy at least 48 hours
* Patient or POA capable of signing informed consent within 48 hours of ICU admission

Exclusion Criteria:

* Past medical history includes cirrhosis
* Active alcohol withdrawal
* Patients taking fluvoxamine prior to admission
* Self-reported hypersensitivity to ramelteon
* Incarcerated patients
* Pregnant patients
* Patients with acute neurological conditions including brain abscess, head bleed, meningitis
* Patients who are transferred from an outside hospital where they have resided for greater than 4 days
* Non-English speaking patients
* Hearing-impaired patients requiring sign language for communication
* Visually-impaired patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Estimated)
Dates: Start 2023-03-26 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Days alive without delirium or coma in the ICU | 14 days
  joint modeling approach taking account recurrence and terminating events

SECONDARY OUTCOMES:
Mean daily Confusion Assessment Method -7 CAM-ICU-7 score | 14 days
  Mean CAM-ICU-7 score
Incidence of delirium, as defined by a positive CAM-ICU-7 | 14 days
  Incidence
Mortality at 14 days from randomization or hospital discharge | 14 days
  Mortality
Duration of delirium, defined as number of days CAM-ICU positive | 14 days
  Duration
ICU length of stay | 14 days
  LOS

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Johnson, MD, Principal Investigator — Centennial Medical Center
Locations (1):
- Centennial Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No